CLINICAL TRIAL: NCT00229853
Title: Thoracoscopic Vascular Rings Chart Review
Status: Terminated | Type: Observational
Why Stopped: sufficient data gathered to support hypothesis
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 04-069
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Cardiovascular Abnormalities
Keywords: Children's Healthcare of Atlanta; pediatric; Thoracoscopic Vascular ring; diverticulopexy; Vascular Ring Division
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to review the use of diverticulopexy, and collect data regarding the ease of the procedure and the overall outcome.

DETAILED DESCRIPTION:
In addition to dividing the vascular ring, some surgeons stress the importance of performing a diverticulopexy (an additional stitch which holds the ring open and prevents recurrence). This is a difficult step to perform through the thoracoscope.

We plan to review the use of this step, the diverticulopexy, and collect data regarding the ease of the procedure and the overall outcome. Once we have accomplished this, we hope to present our initial results of this new procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing vascular ring division at Children's Healthcare of Atlanta at Egleston Hospital between 2001 and 2004

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: retro chart review
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2004-08; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States